CLINICAL TRIAL: NCT02100904
Title: Uterine Leiomyoma Treatment With Radiofrequency Ablation (ULTRA) Registry
Acronym: ULTRA Registry
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 14-13325
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Uterine Fibroids
Keywords: Fibroids; Radiofrequency ablation; Myomectomy
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Women undergoing radiofrequency ablation.: Most women (75%) in the trial will be in the group who receive treatment with radiofrequency ablation (Acessa).
  Interventions: Procedure: Radiofrequency ablation of fibroids
- Women undergoing myomectomy: About 25% of women in the trial will be in the group who receive treatment with myomectomy.
  Interventions: Procedure: Myomectomy of fibroids

INTERVENTIONS:
Procedure: Radiofrequency ablation of fibroids
  Groups: Women undergoing radiofrequency ablation.
Procedure: Myomectomy of fibroids
  Groups: Women undergoing myomectomy

SUMMARY:
The ULTRA Registry is a nationwide observational arm of the ULTRA trial. Data from the ULTRA Registry will be used to evaluate the long-term safety and efficacy of laparoscopic RF ablation (Acessa).

The ULTRA Registry will recruit women age 21 or older who plan to undergo or have undergone laparoscopic RF ablation (Acessa) or myomectomy within the United States. Participants will be recruited through study materials distributed at clinical offices across the country where gynecologists are performing laparoscopic RF ablation (Acessa). Study participants will consent to participate in a 3 year prospective study conducted by UCSF but the fibroid procedure will be performed by the study participants' own gynecologist. We will evaluate changes in fibroid-related symptoms from pre-treatment values to 6, 12, 18, 24, 30, and 36 months after RFA (Acessa). We will determine long-term efficacy of RFA (Acessa) by evaluating the rate of re-treatment for symptomatic fibroids after the RFA (Acessa) procedure versus myomectomy. Participants will be asked for permission to review their medical records to assess surgical and pregnancy outcomes.

UC San Francisco will have oversight of all scientific and administrative aspects of the study. All study data will be stored securely in a HIPAA compliant, secure database monitored by the UC San Francisco Coordinating Center.

ELIGIBILITY:
Inclusion Criteria:

* Planning to undergo or have undergone* RF ablation (Acessa) or myomectomy (laparoscopic or abdominal) for treatment of uterine fibroids.
* Able to give informed consent
* Speak English or Spanish

  * Women enrolled at contracted clinical sites must enroll prior to their RF ablation treatment

Exclusion Criteria:

* <21 years of age
* Plan to undergo hysteroscopic myomectomy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with uterine fibroids who are planning to undergo or have undergone radiofrequency ablation (Acessa) or myomectomy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2014-05; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Changes in fibroid-related symptoms after the RFA or myomectomy procedure. | Baseline to 3 years
  We will use standard questionnaires for women with fibroids to assess changes in fibroid symptoms including menstrual pattern and flow and overall quality of life.

SECONDARY OUTCOMES:
Rate of re-intervention for recurrent fibroid symptoms following the RFA or myomectomy procedure. | Baseline to 6 weeks
Operative complications | Baseline to 6 weeks
  Operative complications are rare but may include excessive blood loss, uterine or pelvic infection, injury to organs adjacent to uterus such as bowel or bladder.
Pregnancy rate after the RFA or myomectomy procedure. | Baseline to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Jacoby, MD, Principal Investigator — University of California, San Francisco
Locations (12):
- United States (12):
  - UC Irvine Medical Center, Irvine, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Dedicated to Women, Dover, Delaware
  - Fibroid and Pelvic Wellness Center of Georgia, Alpharetta, Georgia
  - Gynecology Institute of Chicago, Chicago, Illinois
  - Women's Healthcare Associates of IL, SC, Homewood, Illinois
  - Duke University, Durham, North Carolina
  - Tassone Advanced Gynecology, Austin, Texas
  - UT Southwestern, Dallas, Texas
  - MacArthur Medical Center, Irving, Texas
  - Acacia OBGYN, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rubio EM, Hilton JF, Bent S, Parvataneni R, Oberman E, Saberi NS, Varon S, Schembri M, Waetjen LE, Jacoby VL. Complementary and Alternative Medicine Use Among Women with Symptomatic Uterine Fibroids. J Womens Health (Larchmt). 2023 May;32(5):546-552. doi: 10.1089/jwh.2022.0094. Epub 2023 Apr 6. PMID 37023398
- See also: Fibroid Trials at UCSF — https://clinicaltrials.ucsf.edu/fibroids